CLINICAL TRIAL: NCT04001543
Title: Double-blind Multicenter Phase III Trial Evaluating the Efficacy of an Oral Immunomodulatory Nutrient on Survival During Postoperative Concomitant Chemoradiotherapy in Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Efficacy of an Oral Immunomodulatory Nutrient on Survival During Postoperative Concomitant Chemoradiotherapy in Head and Neck Cancer
Acronym: SIMPA01
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICM-URC 2017/21; GORTEC 2017-02 (Registry Identifier: GORTEC); 2018-A00518-47 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-06-06; First posted 2019-06-28 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma (HNSCC); immunomodulatory nutrient; concomitant chemoradiotherapy; survival
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunomodulating oral supplementation (Experimental): The immunomodulating oral supplementation compound (Oral Impact®) contains 334kcal/bag and 18.1g of proteins, as well as immunomodulatory nutrients such as L-Arginine, RNA and omega-3.
  Each bag of product containing powder (74g/bag) will be diluted in 250 millilitres of water by the patients and drunk at home. Three doses will be drunk at home by the patients daily, during the 5 days before each chemotherapy cycle.
  Interventions: Dietary Supplement: Immunomodulating oral supplementation
- Sip feed control (Active Comparator): The control has the same formula to that of the Oral Impact®, but not enriched with specific nutrients: it is an isocaloric isonitrogenous control.
  Each bag of product containing powder (74g/bag) will be diluted in 250 millilitres of water by the patients and drunk at home. Three doses will be drunk at home by the patients daily, during the 5 days before each chemotherapy cycle.
  Interventions: Dietary Supplement: Sip feed control

INTERVENTIONS:
Dietary Supplement: Immunomodulating oral supplementation — Per os administration, 3 times / day, 5 days before each cycle of chemotherapy.
  Arms: Immunomodulating oral supplementation
Dietary Supplement: Sip feed control — Per os administration, 3 times / day, 5 days before each cycle of chemotherapy.
  Arms: Sip feed control

SUMMARY:
The investigators designed a prospective randomized double-blind trial to determine if the oral immunomodulating formula could improve the disease-free survival rate in high-risk locally-advanced head and neck Squamous Cell Carcinoma patients treated with Chemoradiotherapy.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy on disease-free survival of a formula enriched with L-arginine, omega-3 fatty acids, and ribonucleic acids, taken for 5 days before each cycle of chemotherapy, in patients with high-risk locally-advanced HNSCC treated with postoperative concomitant chemoradiotherapy (CRT).

This study is a national, multicentric double blinded, randomised phase III trial. A total of 306 patients (102 patients in group control vs 204 patients in group Oral Impact®) will be required including 10% of lost-to-follow-up patients.

An immunomodulating oral supplementation compound (Oral Impact®) is compared to an isocaloric isonitrogenous control. The compound to be assessed contains 334kcal/bag and 18.1g of proteins, as well as immunomodulatory nutrients such as L-Arginine, RNA and omega-3. The control has the same formula to that of the Oral Impact®, but not enriched with specific nutrients. Each patient has to take Oral Impact® or a sip feed control during 5 days before each cycle of chemotherapy.

DFS will be measured from the time of randomization to the time of the first evidence of progression (local, regional, metastatic, or second primary) or death from any cause. Patients alive without carcinologic event were censored at last follow-up date.

Patients treated with postoperative CRT are expected to have a 2-year DFS rate of 60% without specific diet (pControl).

Including a ratio 1:2, an expected recruitment of 90 patients per year, the current study will require 131 events to detect an absolute improvement of 15% (HR=0.56, pExperimental=75%) with 0.90 statistical power using a two-sided test and a significance level of 0.05.

A total of 306 patients (102 vs 204) will be required including 10% of lost of follow-up patients.

The inclusion period would be 4 years, for an expected total duration of study about 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Surgically resected primary squamous cell carcinomas (HNSCC) of the hypopharynx, oropharynx, larynx and oral cavity with pathological stage pT1-2 pN+ (pathological stage 1 ou 2 with node) or pT3-4 any pN (pathological stage 3 ou 4 with or without node) (UICC 7th edition, 2010),
* Postoperative concomitant CRT based on radiotherapy and on cisplatinum, 3 cycles, 100mg/m² by cycle,
* Patients who undergone macroscopically complete resection,
* High-risk characteristics patients with one or more following criteria: such as invasion of two or more regional lymph nodes, extracapsular extension of nodal disease or microscopically-involved mucosal margins of resection, perineural involvement, vascular tumor embolism,
* WHO (World Health Organization) performance status 0, 1 or 2,
* Age: 18 years old up to 75 years old including,

Exclusion Criteria:

* Nasopharyngeal, paranasal sinuses, nasal cavity tumours or thyroid cancers
* Sepsis at baseline
* Distant metastasis
* Other immunomodulating diets in the last month before inclusion
* Parenteral nutrition at baseline
* History of hypersensitivity and/or allergy to any component of Oral Impact ®
* Patients with history of malignancies who are not disease-free for more than 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | From date of randomization until the date of the first documented progression (local, regional, metastatic) or date of death from any cause, whichever came first, assessed up to 2 years.
  2-years DFS rate

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization until the date of death from any cause, assessed up to 3 years.
  OS at 1, 2 and 3 years
Rate of drug compliance | up to 45 days
  the compliance is defined as the taking of more than 75 % of study product prescription
Adverse events rate | until 3 months after radiotherapy
  graded based on NCI-CTCAE v4.03
Quality of life by using the general quality of life questionnaire about cancer (QLQ-C30). | Quality of life will be assessed up to 2 years after the last day of radiotherapy.
  The EORTC QLQ-C30 uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Quality of life by using the specific quality of life questionnaire about head and neck cancer (HN35) | Quality of life will be assessed up to 2 years after the last day of radiotherapy.
  The EORTC HN35 uses a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
Cachexia | Cachexia will be assessed up to 3 years after the last day of radiotherapy.
  Cachexia will be evaluated with weight (in kilograms)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SENESSE, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (2):
- France (2):
  - Centre Léon Bérard, Lyon
  - Institut du Cancer de Montpellier, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Background] Bernier J, Domenge C, Ozsahin M, Matuszewska K, Lefebvre JL, Greiner RH, Giralt J, Maingon P, Rolland F, Bolla M, Cognetti F, Bourhis J, Kirkpatrick A, van Glabbeke M; European Organization for Research and Treatment of Cancer Trial 22931. Postoperative irradiation with or without concomitant chemotherapy for locally advanced head and neck cancer. N Engl J Med. 2004 May 6;350(19):1945-52. doi: 10.1056/NEJMoa032641. PMID 15128894
- [Background] Machon C, Thezenas S, Dupuy AM, Assenat E, Michel F, Mas E, Senesse P, Cristol JP. Immunonutrition before and during radiochemotherapy: improvement of inflammatory parameters in head and neck cancer patients. Support Care Cancer. 2012 Dec;20(12):3129-35. doi: 10.1007/s00520-012-1444-5. Epub 2012 Mar 28. PMID 22453793
- [Background] Vasson MP, Talvas J, Perche O, Dillies AF, Bachmann P, Pezet D, Achim AC, Pommier P, Racadot S, Weber A, Ramdani M, Kwiatkowski F, Bouteloup C. Immunonutrition improves functional capacities in head and neck and esophageal cancer patients undergoing radiochemotherapy: a randomized clinical trial. Clin Nutr. 2014 Apr;33(2):204-10. doi: 10.1016/j.clnu.2013.06.008. Epub 2013 Jun 20. PMID 23849811
- [Background] De Geest S, Sabate E. Adherence to long-term therapies: evidence for action. Eur J Cardiovasc Nurs. 2003 Dec;2(4):323. doi: 10.1016/S1474-5151(03)00091-4. No abstract available. PMID 14667488